CLINICAL TRIAL: NCT04489901
Title: The Effect of Olive Oil on Striae Gravidarum in Primiparous Women: A Randomized Controlled Clinical Trial
Brief Title: Stria Gravidarum and Olive Oil for Pregnancy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayca Solt Kirca (Other)
Responsible Party: Sponsor-Investigator, Ayca Solt Kirca, Assistant Professor, Kırklareli University
Organization: Kırklareli University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KırklareliAS
Record Dates: First submitted 2020-07-15; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Striae Gravidarum; Pregnancy Related
Keywords: Striae Gravidarum; primipara women; pregnancy; Olive oil
MeSH Terms: conditions — Striae Distensae | interventions — Olive Oil

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant, Care Provider
Masking Description: This study was a randomized controlled clinical trial. To avoid bias, an impartial midwife who was working in the outpatient clinic on the day the data were collected and was not among the researchers asked each participant to select one of two closed envelopes that included the letters A (experimental group) or B (control group). The pregnant women were assigned to the experimental and control groups depending on the letter in the envelope they chose. Then, the researcher registered the participants in the experimental and control groups on a list. The obstetrician and pregnant women were informed about the procedure, but the obstetrician did not know which procedure would be applied to which pregnant woman. The pregnant women did not know why olive oil was being used. The participating women signed an informed consent form knowing that they could withdraw from the study at any time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extra Virgin Olivei oil group (Experimental): The women in the experimental (olive oil) group were asked to apply 10 cc (4 tablespoons) of extra virgin olive oil to the entire abdomen by hand without massaging twice a day in the morning and evening.
  Interventions: Other: Olive oil
- Control group (No Intervention): The women in the control group did not undergo any intervention.

INTERVENTIONS:
Other: Olive oil — To apply 10 cc (4 tablespoons) of extra virgin olive oil to the entire abdomen by hand without massaging twice a day in the morning and evening.
  Arms: Extra Virgin Olivei oil group

SUMMARY:
The aim of this study was to investigate the clinical efficacy of olive oil on the severity and progression of striae gravidarum. This randomized controlled clinical trial included 156 primipara women who were early third trimester. They were randomly allocated into two groups: an experimental group and a control group. Women in the experimental group applied olive oil to their abdomen twice a day in the morning and evening. The control group had no intervention.

DETAILED DESCRIPTION:
The development of striae is one of the most common skin changes in pregnancy. The aim of this study was to investigate the clinical efficacy of olive oil on the severity and progression of striae gravidarum.

This randomized controlled clinical trial included 156 primipara women who were early third trimester. They were randomly allocated into two groups: an experimental group and a control group. Women in the experimental group applied olive oil to their abdomen twice a day in the morning and evening. The control group had no intervention.Data were collected using maternal information form, Fitzpatrick Skin Type Scale and Davey's Severity Score.

ELIGIBILITY:
Inclusion Criteria:

* being in the age group of 20-30 years, early third trimester (being at the 28th week of gestation), having a singleton pregnancy, being primiparous, and volunteering to participate in the study.

Exclusion Criteria:

* having a chronic disease (such as diabetes or hypertension), having striae (before 28th gestation week), having traces of scar tissue from adolescence, using cortisone cream or another kind of topical cream, having polyhydramnios, having threatened preterm labor or preterm delivery, having any disease of the skin, taking any medication regularly, having a problem preventing communication, using pharmacological or non-pharmacological methods (undergoing pharmacotherapy) to reduce nausea, and undergoing psychiatric treatment (psychotherapy).

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy
Enrollment: 156 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Prevent the severity and progression of SG | All the participating women were followed-up from the 28th week of gestation to the 37th week of gestation.
  The participants completed the Maternal Information Forms through face-to-face interviews with an unbiased midwife who was working in the outpatient clinic on the day the data were collected.The women in the experimental group were asked to apply 10 cc (4 tablespoons) of extra virgin olive oil to the entire abdomen by hand without massaging twice a day in the morning and evening. The control group did not undergo any intervention. The women were called via telephone by the researcher once a week and asked whether they were performing the application. Women who were not applying the olive oil or who were using other medicines or creams (at least three days a week) were excluded from the study. The women in the control group were asked whether they were performing any applications. Those who were applying any products were also excluded. The striae was evaluated all groups at 37 weeks of gestation based on the Fitzpatrick Skin Type Scale and Davey's Severity Score by obstetrician.
Maternal information form | All the participating women were followed-up from the 28th week of gestation to the 37th week of gestation.
  The Maternal Information Form was used to select whether pregnant women met the study.This form, which was developed by the researchers in line with knowledge of the literature, included 30 items questioning the participants' sociodemographic ch criteria.
The Fitzpatrick Skin Type Scale | All the participating women were followed-up from the 28th week of gestation to the 37th week of gestation.
  The Fitzpatrick Skin Type Scale was developed by Fitzpatrick in 1975 to classify skin type.This scale uses genetic structure, eye color, reaction to sunlight to assign a skin type. According to the scale, the skin types vary from the extremely sensitive type, which always burns and does not tan, to the sun-resistant type, which is darkly pigmen and response to sunlight.
Davey's Severity Score | All the participating women were followed-up from the 28th week of gestation to the 37th week of gestation.
  Davey's Severity Score is a scoring method developed by Davey in 1972 to measure the severity of SG.It divides the abdomen into four equal quadrants. Each quadrant is rated as "0" for clean skin, "1" for moderate striae, and "2" for multiple striae. Accordingly, the total score ranges from 0 to 8.

CONTACTS AND LOCATIONS:
Overall Officials: AYCA S KIRCA, Phd, Study Director — Kırklareli University
Locations (2):
- Turkey (Türkiye) (2):
  - Medipol University, Istanbul
  - Kırklareli University, Kırklareli

IPD SHARING:
Plan to Share IPD: Yes
The study will be accessible to everyone after publication in the journal
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data is available now
Access Criteria: The study will be accessible to everyone after publication in the journal

REFERENCES:
- [Derived] Solt Kirca A, Kanza Gul D. Effects of Olive Oil on Striae Gravidarum in Primiparous Women: A Randomized Controlled Clinical Study. Altern Ther Health Med. 2022 May;28(4):34-39. PMID 34559686